CLINICAL TRIAL: NCT04327687
Title: Remote Ischemic Conditioning AS Adjuvant Therapy for Parkinson's Disease: A Prospective, Randomized Controlled Trial
Brief Title: Remote Ischemic Conditioning for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of neurology department, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: k2019-54
Record Dates: First submitted 2020-03-22; First posted 2020-03-31 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Remote ischaemic conditioning
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: a single-blind (outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remote ischemic conditioning (Experimental): remote ischemic conditioning is a physical strategy performed by an electric auto-control device with cuffs placed on bilateral arms: five cycles of 5-min inflation and 5-min deflation one or two times per day. The duration of the treatment is six months.
  Interventions: Device: Remote ischaemic conditioning; Other: conventional therapy
- conventional therapy (Active Comparator): conventional therapy
  Interventions: Other: conventional therapy

INTERVENTIONS:
Device: Remote ischaemic conditioning — 5 cycles of 5 minutes of upper limb ischaemia followed by 5 minutes of reperfusion. This will be delivered using a manual sphygmomanometer applied to the upper arm and activated to go through 5 such cycles automatically. The blood pressure cuff in the active treatment arm will inflate to 200 mmHg. RIC will be completed 1-2 times per day for six months.
  Arms: remote ischemic conditioning
Other: conventional therapy — conventional therapy

SUMMARY:
The purpose is to evaluate feasibility and efficacy of Remote Ischemic Conditioning(RIC) as adjuvant therapy for Parkinson's Disease(PD). Sixty patients will be randomized into 2groups: RIC group receiving Remote Ischemic Conditioning except conventional therapy（n=30）and control group with conventional therapy (n=30).

DETAILED DESCRIPTION:
Remote ischaemic conditioning (RIC) is a procedure whereby ischaemia is induced to a limb for short periods of time by inflating pressure cuffs around arms to above systolic pressures (mmHg). This procedure induce neurohormonal, systemic or vascular changes in the body. Such changes often result in improved collateralisation of blood supply to various areas of the body, as well as improved efficiencies of cellular metabolism. RIC has been shown to improve outcomes in patients with heart attacks, strokes, but is not investigated for PD. We argue that RIC may exert neuroprotective effect on PD due to its multiple mechanisms. The aim of the study is to evaluate the impact of RIC on long term outcomes in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 - 70 years;
* diagnosed with idiopathic PD;
* a rating of 1-3 on the Hoehn and Yahr Scale;
* On optimized dopaminergic therapy for 4 weeks prior to enrollment;
* Be able to complete the research scale evaluation;
* sign informed consent.

Exclusion Criteria:

* Atypical Parkinsonism or other significant brain conditions such as a stroke;
* Significant mental disease or psychosis;
* History or presence of significant peripheral vascular disease in the upper limbs;
* Presence of skin ulceration to the arms;
* Deep Brain Stimulation ( DBS);
* Taking part in another clinical trial of an investigational medicinal product;
* Life expectancy less than 1 year due to Severe medical disease;
* other reasons that are unsuitable for the trial in the investigator's opinion.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Unified Parkinson's disease Rating Scale - Session III | 24weeks
  The Unified Parkinson´s Disease Rating Scale Part Ⅲ is an accepted and validated scale for the assessment of motor function in Parkinson´s disease. Each of the 27 sub-items in the UPDRS III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities. The total scores therefore ranges from 0 (Best score possible) to 108 (Worst score possible).

SECONDARY OUTCOMES:
Change in Unified Parkinson's disease Rating Scale - Session III | 12 weeks, 48 weeks
  The Unified Parkinson´s Disease Rating Scale Part Ⅲ is an accepted and validated scale for the assessment of motor function in Parkinson´s disease. Each of the 27 sub-items in the UPDRS III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities. The total scores therefore ranges from 0 (Best score possible) to 108 (Worst score possible).
Changes on Depression | 12 weeks, 24weeks, 48 weeks
  Assessment with Beck's depression inventory (BDI) .
Changes on Cognitive function | 12 weeks, 24weeks, 48 weeks
  Rating with Montreal Cognitive Assessment (MOCA)
Changes on quality of life | 12 weeks, 24weeks, 48 weeks
  It will be evaluated through the Parkinson Disease Questionnaire (PDQ-39).
Levodopa Equivalent Dose | 12 weeks, 24weeks, 48 weeks
  Assessment with Research Team
frequency of adverse events | From screening up to 48 weeks
  Adverse events to evaluate the safety and tolerability of Remote ischaemic conditioning

CONTACTS AND LOCATIONS:
Overall Officials: Chen Hui-Sheng, Study Chair — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: No